CLINICAL TRIAL: NCT06448325
Title: RIFRA - Re-fracture Risk Prediction in Patients With Fragility Fracture: Score Development and Validation
Brief Title: Fragility Re-fractures Prediction Score
Acronym: RIFRA
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: RIFRA
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Osteoporosis Risk
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hip arthroplasty — Surgical treatment of the hip after osteoporosis fracture. The focus of the study is the prediction of further fractures (and therefore further surgical procedures) after the first one.

SUMMARY:
Fragility fractures increase among elderly patients worldwide, representing a global burden in terms of disability and care expenditure.

Osteoporosis is asymptomatic up to the moment in which a first fracture occurs, reason why it is often underdiagnosed. Even after that, further fractures do occurr, as osteoporosis is often untreated. Several programs have been introduced worldwide to prevent secondary fractures among the population at risk (e.g., International Osteoporosis Foundation's Capture the Fracture), and several risk factors are being investigated to generate a predictive score. However, accurate validation is needed to make these scores reliable.

In this retrospective observational study, we aim to validate a predictive score trained on a population of elderly patients with a cohort of patients who underwent hip fracture surgery in a high-volume orthopedic center in the Region of Lombardy.

ELIGIBILITY:
Inclusion Criteria:

* People who underwent total or partial hip replacement (ICD 9 CM 81.51, 81.52) in five years (2013-2017) at the hospital for a compound fracture of the hip (ICD 9 CM 820, 820.01-820.09).

Exclusion Criteria:

* People undergoing the same intervention for other reasons (e.g. pathological fracture, ICD 9 CM 733.14).

ICD 9 CM stands for International Classification of Disease, 9th Revision, Clinical Modification.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 or more, of all sexes.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Age, sex, disease name and body mass index (weight in kg and height in m will be combined to report BMI in kg/m^2) | Baseline: the outcomes are assessed before surgery
  Patient characteristics and comorbidities associated with a fragility fracture of the hip

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided